CLINICAL TRIAL: NCT00238394
Title: A Phase II Study of AZD2171 in Patients With Locally Advanced or Metastatic Hepatocellular Carcinoma
Brief Title: Cediranib Maleate in Treating Patients With Locally Advanced or Metastatic Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01822; N044J; CDR0000446081; NCCTG-N044J; U10CA025224 (NIH)
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — cediranib

ARMS (1):
- Treatment (cediranib maleate) (Experimental): Patients receive oral AZD2171 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a CR receive 2 additional courses beyond CR. Patients experiencing disease progression within 5 years after completion of study treatment may receive additional courses of study treatment.
  Interventions: Drug: cediranib maleate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cediranib maleate — Given orally
  Other Names: AZD2171; Recentin
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
AZD2171 (cediranib maleate) may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. This phase II trial is studying how well AZD2171 works in treating patients with locally advanced or metastatic liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the 6-month survival of patients with locally advanced or metastatic hepatocellular carcinoma treated with AZD2171.

SECONDARY OBJECTIVES I. Determine tumor response and time to progression in patients treated with this drug.

II. Determine the toxicity of this drug in these patients. III. Correlate biological markers with response in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral AZD2171 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 additional courses beyond CR. Patients experiencing disease progression within 5 years after completion of study treatment may receive additional courses of study treatment.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 4 years.

PROJECTED ACCRUAL: A total of 20-44 patients will be accrued for this study within 22 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed hepatocellular carcinoma

  * Locally advanced or metastatic disease
  * Not amenable to treatment with surgery or orthotopic liver transplantation
* Measurable or non-measurable disease

  * Measurable disease is defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* Evidence of disease progression by imaging on serial exams or biochemical evidence of a rising alpha fetoprotein on serial testing
* No history of brain metastases other than locally treatable CNS lesions (i.e., lesions treatable with surgery or radiosurgery)

  * Patients with locally treatable CNS disease eligible provided they were previously treated and had no evidence of CNS progression for ≥ 4 weeks after completion of treatment
* No fibrolamellar hepatocellular carcinoma or mixed cholangiocarcinoma/hepatocellular carcinoma
* Performance status - ECOG 0-1
* Absolute neutrophil count ≥ 1,200/mm^3
* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 10.0 g/dL
* Bilirubin ≤ 3 times upper limit of normal (ULN)
* AST ≤ 5 times ULN
* Alkaline phosphatase ≤ 5 times ULN
* Urine protein < 1+ by urine dip stick OR proteinuria < 1 gm/24-hour collection
* QTc prolongation ≤ 500 msec
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No uncontrolled blood pressure, defined as systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 100 mm Hg
* No significant ECG abnormality within the past 14 days
* No New York Heart Association class III or IV disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No history of allergic reaction to compounds of similar chemical or biological composition to AZD2171
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study participation
* No other uncontrolled illness
* More than 4 weeks since prior biologic therapy
* More than 4 weeks since prior and no concurrent immunotherapy
* No colony-stimulating factors during the first course of study treatment
* At least 6 weeks since prior chemoembolization

  * Patients must have evidence of disease progression or new metastases after prior chemoembolization
* No prior systemic chemotherapy for this cancer
* No other concurrent chemotherapy
* More than 4 weeks since prior hormonal therapy
* See Disease Characteristics
* At least 6 weeks since prior radiofrequency ablation or other local ablative therapy

  * Patients must have evidence of disease progression or new metastases after prior radiofrequency ablation or other local ablative therapy
* No prior external beam radiotherapy to the primary site
* No prior radiotherapy to ≥ 25% of the bone marrow
* No concurrent radiotherapy
* See Disease Characteristics
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent drugs or biologics with proarrhythmic potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-12; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Survival after 6 months of treatment | 6 months
  Will be estimated by the proportion of patients surviving more than 6 months. Ninety-five percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.
Time to disease progression | From registration to documentation of disease progression, assessed up to 5 years
  Will be estimated using the method of Kaplan-Meier.

SECONDARY OUTCOMES:
Confirmed tumor response is defined to be a CR or PR noted as the objective status on 2 consecutive evaluations at least 4 weeks apart | Up to 5 years
Laboratory measures | Up to 5 years
  Descriptive statistics will be computed for the laboratory measures, including frequency and Cox proportional hazards modeling.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Alberts, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States